CLINICAL TRIAL: NCT04213105
Title: A Randomized, Double-blind and Parallel Group Study to Compare the Pharmacokinetic, Safety and Pharmacodynamic of QL1206 and Prolia® in Healthy Adults
Brief Title: Comparing of the Pharmacokinetic, Safety and Pharmacodynamic of QL1206 and Prolia® in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QL1206-002
Record Dates: First submitted 2019-12-10; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Healthy People
MeSH Terms: interventions — QL1206; Denosumab

STUDY DESIGN:
Intervention Model Description: randomized、double-blind、parallel-group、positive control
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1206 (Experimental): QL1206 injection (60mg) by subcutaneous injection once on the first day
  Interventions: Drug: QL1206
- Prolia® (Active Comparator): Prolia® injection (120mg) by subcutaneous injection once on the first day
  Interventions: Drug: Prolia®

INTERVENTIONS:
Drug: QL1206 — subcutaneous injection of 60 mg (1ml) only once,on the first day.
  Arms: QL1206
Drug: Prolia® — subcutaneous injection of 60 mg (1ml)only once,on the first day
  Other Names: Denosumab Injection
  Arms: Prolia®

SUMMARY:
A randomized, double-blind and parallel group study to compare the pharmacokinetic, safety and pharmacodynamic of QL1206 and Prolia® in healthy adults

DETAILED DESCRIPTION:
This is a phase I,single center, randomized, double-blind and parallel group clinical trial . The primary objective is to assess the pharmacokinetic similarity of single and subcutaneous injections of QL1206 or Prolia® in healthy volunteers. The secondary objective are to assess the Clinical safety and immunogenicity similarity of single and subcutaneous injections of QL1206 or Prolia® in healthy volunteers. Meanwhile，observing the pharmacodynamic similarities of QL1206 or Prolia® preliminarily. Subjects would receive a single 60mg（1ml） of QL1206 or through subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form and fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the test plan requirements;
* Aged ≥18 years or ≤50 years, male or female (including the boundary value);
* Agree to take effective contraceptive measures throughout the study period (including not limited to: hormonal drugs of pregnancy, physical contraception, surgery, abstinence, etc., until at least 6 months after the last study is administered;
* Clinical laboratory examination, chest X-ray, abdominal B-ultrasound, electrocardiogram, physical examination, vital signs and various examinations are normal or abnormal without clinical significance

Exclusion Criteria:

* Occurred or suffering from osteomyelitis or ONJ (mandibular necrosis) previously.
* Serum calcium levels are outside the normal range of the laboratory, or the subject uses calcium supplements in the screening period.
* The dental or jaw disease that is active, requiring oral surgery; or planned for invasive dental surgery during the study; or dental or oral surgery wounds have not healed;
* Subject has viral hepatitis (including hepatitis B and hepatitis C), AIDS antibodies, and Treponema pallidum antibodies;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-t ) | 134 day
  Area under the plasma concentration-time curve (AUC0-t ) from 0 o'clock to the last measurable concentration acquisition time t.
maximum plasma concentration(Cmax) | 134 day
  the maximum plasma concentration of QL1206/Prolia from 0 o'clock to the last measurable concentration acquisition time t.

SECONDARY OUTCOMES:
Adverse events(AE) | 134 day
  The adverse medical events that occur after the clinical trial subjects receive the test drug do not necessarily have a causal relationship with the treatment.
serum CTX1 | 134 day
  CTX1 is a serum type I collagen C-terminal peptide to detect the bone metastasis. the secondary outcome measures the percent change in serum CTX1 throughout the study from baseline to 134 day

CONTACTS AND LOCATIONS:
Overall Officials: yanhua DING, Professor, Principal Investigator — The First Affiliated Hospital of Jilin University
Locations (1):
- The First Affiliated Hospital of Jilin University, Changchun, Jilin, China